CLINICAL TRIAL: NCT00002952
Title: Phase I/II Study of Immunization With MAGE-3 Peptide-Pulsed Autologous PBMC Plus rhIL-12 in Patients With Metastatic Melanoma
Brief Title: Vaccine Therapy and Interleukin-12 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9018; UCCRC-9018; UCCRC-8381; NCI-G97-1162
Record Dates: First submitted 1999-11-01; First posted 2004-04-22 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — MART-1 Antigen; MAGEA3 protein, human; Interleukin-12 Subunit p35

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): Melan-A peptide loaded PBMCs (sc, q3wk x 3), rhIL-12 (4 mcg, sc, days 1, 3 and 5 of every 3 wk cycle)
  Interventions: Biological: MART-1 antigen; Biological: recombinant MAGE-3.1 antigen; Biological: recombinant interleukin-12

INTERVENTIONS:
Biological: MART-1 antigen — Melan-A peptide loaded PBMCs (sc, q3wk x 3)
Biological: recombinant MAGE-3.1 antigen
  Other Names: Melan-A peptide loaded PBMCs (sc, q3wk x 3)
Biological: recombinant interleukin-12 — rhIL-12 (4 mcg, sc, days 1, 3 and 5 of every 3 wk cycle)

SUMMARY:
RATIONALE: Vaccines made from a tumor antigen gene may make the body build an immune response to kill tumor cells. Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cell to kill melanoma cells. Combining vaccine therapy with interleukin-12 may kill more melanoma cells.

PURPOSE: Phase I/II trial to study the effectiveness of vaccine therapy plus interleukin-12 in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and maximum tolerated dose level of the vaccine consisting of MAGE-3 or Melan-A (human tumor antigen genes) peptide-pulsed autologous peripheral blood mononuclear cells plus interleukin-12. II. Determine if the procedure results in successful immunization. III. Assess the response of the tumor to the vaccine.

OUTLINE: This is an open label, nonrandomized, single institution study. Patients receive 3 initial courses of treatment consisting of 21 days each. Treatment consists of an immunization with MAGE-3 or Melan-A peptide-loaded autologous PBMC and interleukin-12 (IL-12) on the first day, IL-12 on days 3 and 5, and 16 days of rest. The first cohort is not administered IL-12 and the next cohorts are given escalating doses of IL-12. The Phase II dose will be one dose level below the MTD. Patients who have a tumor remission response or stable disease may continue treatment for up to one year. Phase I completed as of 04/1999. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 34 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic melanoma Patient must express HLA-A2 (a human leukocyte antigen) Tumor must express MAGE-3 or Melan-A by polymerase chain reaction (PCR) analysis No untreated brain metastases

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Karnofsky 70%-100% Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin no greater 1.5 times upper limit of normal (ULN) SGPT no greater than 2 times ULN Renal: Calcium no greater than 11 mg/dL Creatinine no greater than 1.5 times ULN Cardiovascular: No significant cardiovascular disease or cardiac arrhythmia requiring medical intervention Other: Hepatitis B surface antigen negative HIV negative No serious concurrent infection No clinically significant autoimmune disease No active gastrointestinal bleeding or uncontrolled peptic ulcer disease No history of inflammatory bowel disease No psychiatric illness that may interfere with compliance in study Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunosuppressive drugs At least 4 weeks since biologic therapy Chemotherapy: At least 2 weeks since chemotherapy Endocrine therapy: No concurrent systemic corticosteroids (except physiologic replacement doses) Radiotherapy: At least 2 weeks since radiotherapy Surgery: At least 2 weeks since surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1997-01; Primary Completion 2002-08 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Clinical Response Rate | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F. Gajewski, MD, PhD, Study Chair — University of Chicago
Locations (1):
- University of Chicago Cancer Research Center, Chicago, Illinois, United States